CLINICAL TRIAL: NCT05643911
Title: Effects of High-flow Oxygen Therapy and Non-invasive Ventilation on Lung Volumes and on Upper Airway in Hypoxemic Critical Care Patients: a Physiological Randomized Controlled Trial
Brief Title: Effects of High-flow Oxygen Therapy and Non-invasive Ventilation on Lung Volumes and on Upper Airway
Acronym: HONIVAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL22_0510
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure
Keywords: intensive care; non-invasive ventilation; high-flow nasal oxygen therapy; hypoxemic respiratory failure; upper airway
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Hight-flow oxygen therapy) (Experimental): In the HFNC group, patients will receive HFNC oxygen therapy for 20 minutes. Oxygen will be passed through a heated humidifier and continuously delivered through medium or large nasal cannulas (OptiflowTM, Fisher and Paykel Healthcare) depending on patient anatomy, with a gas flow of 50 litres per minute and the FiO2 will be adjusted to maintain a SpO2 between 95% and 98%.
  Interventions: Procedure: HFNC
- Non-invasive ventilation (NIV) (Active Comparator): In the NIV Group, patients will receive NIV for 20 minutes delivered with a naso-buccal or face mask according to the patient's tolerance. The pressure-support level will be adjusted with the aim of an expired tidal volume of 6 to 8 ml per kilogram of predicted body weight, with a positive end-expiratory pressure (PEEP) of 5 cmH2O. The FiO2 will be adjusted to maintain a SpO2 between 95% and 98%.
  Interventions: Procedure: NIV

INTERVENTIONS:
Procedure: HFNC — In the HFNC group, patients will receive HFNC oxygen therapy for 20 minutes.
  Arms: HFNC (Hight-flow oxygen therapy)
Procedure: NIV — Patients will receive NIV for 20 minutes delivered with a naso-buccal or face mask according to the patient's tolerance.
  Arms: Non-invasive ventilation (NIV)

SUMMARY:
Respiratory failure is the most frequent organ failure and cause for admission in the Intensive Care Unit (ICU) . It is a severe complication with an ICU mortality ranged from 31% to 33%. Symptomatic treatment of hypoxemic respiratory failure is a controversial topic with different options: 1) standard oxygen therapy, 2) high flow nasal cannula oxygen therapy (HFNC) and 3) non-invasive ventilation (NIV).

The aim of the study is to compare HFNC versus NIV ventilation using CT scan. The hypothesis of this study is that in hypoxemic critically ill patients, the increase of lung volumes with NIV would be significantly higher than the increase of lung volumes with HFNC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hypoxemia at any time of ICU stay defined as follow: standard oxygen therapy flow ≥ 3L/min to maintain a pulsed oxygen saturation ≥ 95%
* Adult (age ≥ 18 years)
* (2) A CT scan prescribed by the physician in charge of the patient as part of the exploration of the patient's pathology and not as part of a "dedicated" prescription for the study.

Exclusion Criteria:

* NIV contraindication (need for immediate endotracheal intubation and mechanical ventilation; hemodynamic instability defined by systolic blood pressure < 90 mmHg or mean blood pressure < 65 mmHg, use of vasopressors; Glasgow Coma Scale score of 12 points or less)
* History of recent facial trauma not compatible with the use of nasal cannulas
* Pregnancy
* Refusal of study participation
* protected person
* Patient not affiliated to the social security system or not benefiting from such a system
* Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Variation in poorly aerated lung volume | the day of inclusion
  The poorly aerated volume will be measured by CT scan
Variation in non-aereted lung volume | the day of inclusion
  The non-aereted volume will be measured by CT scan

SECONDARY OUTCOMES:
Variation in cross-sectional upper airway area | the day of inclusion
  The variation will be measured by CT-scan in mm
Variation in normally aerated lung volume | the day of inclusion
  The normally aerated lung volume will be measured by CT scan
Variation in Positive End Expiratory Pressure (PEEP) | the day of inclusion
Variation in Total lung volume | the day of inclusion
  The total lung volume will be measured by CT-scan
Variation in O2 gas exchange | the day of inclusion
  Change in PaO2 in mmHg
Variation in CO2 gas exchange | the day of inclusion
  Change in PaO2 in mmHg
Variation in respiratory rate | the day of inclusion
  Respiratory rate is the number of cycles per minute
Variation in cardiac output (Qc) | the day of inclusion
  the cardiac output is in L/min
Variation in patient comfort | the day of inclusion
  Patient comfort through a numeric rating scale (NRS) from 0 (no discomfort) to 10 (maximum imaginable discomfort)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Montpellier, Saint Eloi, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and institutional review board (IRB) review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Derived] Monet C, Piron L, Pressac M, Molinari N, De Jong A, Guiu B, Jaber S. Study protocol for the HONIVAH trial: a single-centre randomised study assessing high-flow oxygen therapy versus non-invasive ventilation on lung volumes and the upper airway in hypoxemic critically ill patients. BMJ Open. 2025 Sep 16;15(9):e106340. doi: 10.1136/bmjopen-2025-106340. PMID 40962342